CLINICAL TRIAL: NCT00911807
Title: A Randomized, Double-Blind, Clinical Trial to Compare the Safety and Efficacy of Cerebrolysin and Aricept (Donepezil) and a Combination Therapy in Patients With Probable Alzheimer's Disease (AD)
Brief Title: Comparative Study to Test Safety and Efficacy of Neurotrophic and Cholinergic Treatment of Alzheimer's Disease
Acronym: Combi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: acromion GmbH (Industry)
Responsible Party: Dr. Philipp Novak, EBEWE Neuro Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBE-031010
Record Dates: First submitted 2009-04-07; First posted 2009-06-02 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer Disease
Keywords: Clinical Trial, Phase II; Randomized Controlled Trial; Multicenter Study; Cerebrolysin; Donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — cerebrolysin; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cerebrolysin + donepezil (Experimental)
  Interventions: Drug: Cerebrolysin + donepezil
- Cerebrolysin + placebo (Experimental)
  Interventions: Drug: Cerebrolysin + placebo
- Donepezil + placebo (Active Comparator)
  Interventions: Drug: Donepezil + placebo

INTERVENTIONS:
Drug: Cerebrolysin + donepezil — Cerebrolysin (10 ml) was given as IV infusion on five days per week for four consecutive weeks (week 1-4) with repetition of this treatment course (week 13-16) after a two-months treatment free interval, accounting for a total of 40 infusions.
  Donepezil was given PO once daily during the whole study duration (28 weeks). After four weeks the daily dosage was increased from 5 mg to 10 mg.
  Other Names: Brand name for donepezil: Aricept; Brand name for Cerebrolysin: Cerebrolysin
  Arms: Cerebrolysin + donepezil
Drug: Cerebrolysin + placebo — Cerebrolysin (10 ml) was given as IV infusion on five days per week for four consecutive weeks (week 1-4) with repetition of this treatment course (week 13-16) after a two-months treatment free interval, accounting for a total of 40 infusions.
  Placebo for donepezil was given PO once daily during the whole study duration (28 weeks).
  Other Names: Brand name for Cerebrolysin: Cerebrolysin
  Arms: Cerebrolysin + placebo
Drug: Donepezil + placebo — Placebo for Cerebrolysin was given as IV infusion on five days per week for four consecutive weeks (week 1-4) with repetition of this treatment course (week 13-16) after a two-months treatment free interval, accounting for a total of 40 infusions.
  Donepezil was given PO once daily during the whole study duration (28 weeks). After four weeks the daily dosage was increased from 5 mg to 10 mg.
  Other Names: Brand name for donepezil: Aricept
  Arms: Donepezil + placebo

SUMMARY:
The study was performed to compare the safety and efficacy of Cerebrolysin (10 mililiters [ml]), Aricept (10 miligrams [mg]), and a combination of both treatments on cognitive performance and global function in patients with probable Alzheimer's Disease (AD). It should also be assessed if the treatments have a positive effect on activities of daily living and neuropsychiatric symptoms.

Oral treatment with Aricept or Placebo was given once daily throughout the study. Intravenous treatment with Cerebrolysin or Placebo was given once daily for 5 days per week during week 1 to 4 and during week 13 to 16 of the study. During the study patients had six visits at the hospital for evaluation.

DETAILED DESCRIPTION:
Endogenous neurotrophic factors, also called neurotrophins, are signaling molecules in various cellular pathways and allow proper neuronal function, survival and regeneration. Sufficient supply is therefore regarded as a pre-requisite for neuronal maintenance but sudden or chronic pathological changes result in an imbalance of this regulatory system.

Cerebrolysin is a peptide preparation acting in a similar way like endogenous neurotrophic factors. Due to its pleiotropic effects - neuroprotection, neuronal survival, neuroplasticity and neurogenesis -, Cerebrolysin is regarded as potential therapeutic tool in complex diseases like stroke or dementia. In contrast to naturally occurring neurotrophic factors, neuropeptides of Cerebrolysin enter the brain parenchyma by crossing the blood-brain barrier after peripheral (intravenous [IV]) administration.

Another treatment approach for Alzheimer's disease targets the cholinergic system to increase cortical acetylcholine. One of these drugs is the anticholinesterase donepezil (Aricept). However, anticholinesterases seem to provide only symptomatic benefit for a limited period and not to influence the progression of the disease. In view of the different mechanisms of action and clinical profile of Cerebrolysin and Aricept, a combination therapy of both may provide synergistic treatment effects. The combination of a treatment targeting the neurotrophic axis (Cerebrolysin) with a treatment to improve cholinergic neurotransmission (Aricept) can arguably be expected to provide additional benefits to AD patients.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of probable AD (Diagnostic and Statistical Manual of Mental Disorders, 4th revision [DSM-IV], National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association [NINCDS-ADRDA])
* Mini-Mental-State-Examination (MMSE) of 12-25, inclusive
* Modified Hachinski score ≤4
* Computed tomography (CT) or magnetic resonance imaging (MRI) scan within 12 months prior to screening without evidence of infection, infarction, or other focal lesions and without clinical symptoms suggestive of intervening neurological disease. Patients who have had a single, clinically silent lacunar infarct are eligible provided the lacunar infarct is not felt to be responsible for the patient's symptoms, is <1 centimeter (cm) maximal diameter in any dimension, is not present in hippocampus of either hemisphere, head of the left caudate, or the dorsomedial region of the left thalamus. Subjects with scans showing atrophy, ventricular enlargement or mild to moderate white matter changes (involving up to approximately 25% of hemispheric white matter) are eligible if the study is otherwise normal.
* Hamilton Depression Scale score of ≤15
* Adequate visual and auditory acuity to allow neuropsychological testing
* Ability to attempt all sections of the Alzheimer's Disease Assessment Scale Cognitive Subpart (extended version)(ADAS-cog+)
* Good general health without additional diseases expected to interfere with the study
* Normal B12, folic acid, venereal disease research laboratory (VDRL), and thyroid-stimulating hormone (TSH) or without any clinically significant laboratory abnormalities that would be expected to interfere with the study
* Electrocardiogram (ECG) and chest x-ray (if clinically necessary per Investigator) without clinically significant laboratory abnormalities that would be expected to interfere with the study
* Patient is not institutionalized
* Patient is not pregnant, lactating, or of childbearing potential
* Sufficient language skills to complete all testing without assistance of a language interpreter
* Responsible caregiver being present during administration of study drug, monitor the patient's compliance with study procedures and adverse events, and accompany the patient to all clinic visits
* Written informed consent obtained from the patient and caregiver prior to entry into the study

Exclusion criteria

* Any clinically significant laboratory abnormalities on the battery of screening tests
* Patients who in the past have not tolerated treatment with 10 mg Aricept or treatment with a corresponding dose of another cholinesterase inhibitor
* Severe psychotic features, depression, agitation or behavioral problems within the last three months that could lead to difficulty complying with the protocol
* Any significant systemic illness or unstable medical condition that could lead to difficulty complying with the protocol
* Patients who in the Investigator's opinion would not comply with study procedures
* Any significant neurological disease other than Alzheimer's Disease, within the past five years, or with residual effects
* Delusional symptoms are often characteristic of Alzheimer's Disease, but patients with symptoms so pronounced that they warrant an alternative diagnosis are excluded
* History of alcohol or substance abuse or dependence within the past two years (DSM-IV)
* History of schizophrenia (DSM-IV)
* Patients with a history of systemic cancer within the past two years are excluded
* History of myocardial infarction in the past year or unstable or severe cardiovascular disease, including uncontrolled hypertension
* Uncontrolled insulin-requiring diabetes or non-insulin dependent diabetes mellitus (Haemoglobin A1c [HBA1c] > 10.0)
* Use of:

  * systemic corticosteroids for more than one week within three months prior to Baseline (BL)
  * Anti-Parkinsonian agents within two months prior to baseline (BL)
  * Approved or investigational Cholinesterase Inhibitors within 30 days or five half-lives, whichever is longer, prior to BL
  * Memantine or other N-methyl-D-aspartic acid (NMDA) antagonists within 30 days or five half-lives, whichever is longer, prior to BL
  * Treatment with high potency neuroleptics or narcotic analgesics within four weeks prior to BL
  * Cimetidine within four weeks prior to BL
  * Sedatives more frequently than two times per week for sleep within four weeks prior to BL

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ánton X Àlvarez, MD, PhD, Principal Investigator — EuroEspes Biomedical Research Center; Herbert Moessler, PhD, Study Director — EBEWE Pharma
Locations (3):
- Spain (3):
  - EuroEspes Biomedical Research Centre, A Coruña
  - Centro Geriátrico Fuente Salinas, Granada
  - Clínica de Memoria, Málaga

REFERENCES:
- [Derived] Alvarez XA, Cacabelos R, Sampedro C, Couceiro V, Aleixandre M, Vargas M, Linares C, Granizo E, Garcia-Fantini M, Baurecht W, Doppler E, Moessler H. Combination treatment in Alzheimer's disease: results of a randomized, controlled trial with cerebrolysin and donepezil. Curr Alzheimer Res. 2011 Aug;8(5):583-91. doi: 10.2174/156720511796391863. PMID 21679156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 18-OCT-2004 - 29-OCT-2007 Type of location: hospital (La Coruna), institutions specialized on cognitive disorders (Granada, Malaga)
Pre-assignment Details: Patients were excluded from the trial before assignment to groups when not all inclusion criteria were met or when exclusion criteria were applicable.
Period: Overall Study
Arm/Group | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil
Started | 72 | 70 | 75
Completed | 55 | 52 | 52
Not Completed | 17 | 18 | 23
Not completed — Adverse Event | 2 | 1 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Protocol Violation | 6 | 4 | 9
Not completed — Withdrawal by Subject | 8 | 10 | 7
Not completed — Organizational reasons | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil | Total
Number analyzed (Participants) | 72 | 70 | 75 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 9 | 9 | 6 | 24.0
  >=65 years | 63 | 61 | 69 | 193.0
Age Continuous [Mean (Standard Deviation); unit: years] | 74.5 (8.3) | 75.1 (7.6) | 76.0 (7.7) | 75.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 58 | 169.0
  Male | 12 | 19 | 17 | 48.0
Region of Enrollment [Number; unit: participants]
  Spain | 72 | 70 | 75 | 217.0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale Cognitive Subpart (Extended Version) (ADAS-COG+) at Week 28
Description: The ADAS-cog+ is a validated, widely used, 14 item psychometric instrument for testing cognitive functions with increased sensitivity in detecting changes in milder patients compared to the original ADAS-cog. It has a maximum score of 85 with a higher score indicating impairment and was assessed by a qualified neuropsychologist.
Time Frame: baseline and week 28
Population: Analysis was intention to treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil
Number analyzed (Participants) | 67 | 64 | 66
points on a scale | -2.348 (5.993) | -1.711 (7.500) | -1.246 (6.147)
Statistical Analysis 1: Comparison: Cerebrolysin + Donepezil vs Cerebrolysin vs Donepezil; The null-hypothesis stated no differences between the three treatment groups regarding the mean change from baseline in ADAS-cog+ at week 28. A sample size of approximately 60 evaluable patients per treatment arm was estimated to allow for the detection of a significant group difference of two points in ADAS-cog+ week 28 change score (standard deviation [SD] 3.3) between the three groups with a power of > 80% and a probability level of alpha = 0.05 (two-sided); Test type: Superiority or Other; p = 0.6348, ANCOVA — ANCOVA F-test. The study was designed to show significant differences in each of the two primary variables. No adjustment for multiple testing was needed and all tests were done with retention of the full two-sided alpha-level of 0.05; ANCOVA with the week 28 ADAS-cog+ change score as dependent variable and the ADAS-cog+ baseline score as a covariate; Mean Square (Factor Treatment) = 19.59
Statistical Analysis 2: Comparison: Cerebrolysin + Donepezil vs Cerebrolysin; Multiple testing of individual null hypotheses that control for the overall significance level alpha = 0.05 were performed by using the 'closed testing procedure'; Test type: Superiority or Other; p = 0.5830, t-test, 2 sided — No adjustment for multiple testing was needed and all tests were done with retention of the full two-sided alpha-level of 0.05; Comparisons between all pair of means were performed with two-sample t-tests within the ANCOVA model; Mean Difference (Final Values) = -0.630, 95% CI [-2.891 to 1.630]
Statistical Analysis 3: Comparison: Cerebrolysin + Donepezil vs Donepezil; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3434, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Comparisons between all pair of means were performed with two-sample t-tests within the ANCOVA model; Mean Difference (Final Values) = -1.080, 95% CI [-3.324 to 1.163]
Statistical Analysis 4: Comparison: Cerebrolysin vs Donepezil; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6962, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Comparisons between all pair of means were performed with two-sample t-tests within the ANCOVA model; Mean Difference (Final Values) = -0.450, 95% CI [-2.719 to 1.819]

2. Primary Outcome: Clinical Interview-based Impression of Change (CIBIC+) Score
Time Frame: week 28
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline for ADAS-COG+
Time Frame: week 4, 12, 16
Reporting Status: Not Posted

4. Secondary Outcome: ADAS-COG+ Responders
Time Frame: week 4, 12, 16, 28
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline for Original ADAS-COG
Time Frame: week 4, 12, 16, 28
Reporting Status: Not Posted

6. Secondary Outcome: CIBIC+ Score
Time Frame: week 4, 12, 16
Reporting Status: Not Posted

7. Secondary Outcome: CIBIC+ Responders
Time Frame: week 4, 12, 16, 28
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Interview-based Impression of Severity (CIBIS+) Score
Time Frame: week 28
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline for Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL)
Time Frame: week 16, 28
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Total Score for Neuropsychiatric Inventory (NPI)
Time Frame: week 16, 28
Reporting Status: Not Posted

11. Secondary Outcome: Combined Responders, i.e. Response in ADAS-COG+ and CIBIC+
Time Frame: week 4, 12, 16, 28
Reporting Status: Not Posted

12. Secondary Outcome: Adverse Experiences, Vital Signs, Physical and Neurological Examinations, Laboratory Tests (Hematology, Clinical Chemistry , Urinalysis, Electrocardiogram [ECG])
Time Frame: Baseline, week 4, 12, 16, 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 2
Other Adverse Events (participants affected / at risk) | 45 | 40 | 46
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil
Pyrexia (General disorders) | 0/67 (0) | 1/65 (1) | 0/68 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0/67 (0) | 1/65 (1) | 0/68 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/67 (0) | 0/65 (0) | 1/68 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0/67 (0) | 0/65 (0) | 1/68 (1)
Respiratory tract infection (Infections and infestations) | 1/67 (1) | 0/65 (0) | 0/68 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/67 (1) | 0/65 (0) | 0/68 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Cerebrolysin + Donepezil | Cerebrolysin | Donepezil
Dyspepsia (Gastrointestinal disorders) | 5/67 (5) | 5/65 (5) | 7/68 (7)
Agitation (Psychiatric disorders) | 4/67 (4) | 9/65 (9) | 3/68 (3)
Dizziness (Nervous system disorders) | 7/67 (7) | 6/65 (6) | 2/68 (2)
Nasopharyngitis (Infections and infestations) | 4/67 (4) | 5/65 (5) | 6/68 (6)
Dysthymic disorder (Psychiatric disorders) | 7/67 (7) | 3/65 (3) | 4/68 (4)
Diarrhoea (Gastrointestinal disorders) | 5/67 (5) | 2/65 (2) | 6/68 (6)
Anorexia (Metabolism and nutrition disorders) | 4/67 (4) | 5/65 (5) | 3/68 (3)
Anxiety (Psychiatric disorders) | 3/67 (3) | 3/65 (3) | 6/68 (6)
Confusional state (Psychiatric disorders) | 3/67 (3) | 5/65 (5) | 4/68 (4)
Nausea (Gastrointestinal disorders) | 5/67 (5) | 1/65 (1) | 6/68 (6)
Headache (Nervous system disorders) | 5/67 (5) | 4/65 (4) | 2/68 (2)
Insomnia (Psychiatric disorders) | 3/67 (3) | 5/65 (5) | 3/68 (3)
Urinary tract infection (Infections and infestations) | 4/67 (4) | 4/65 (4) | 3/68 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No